CLINICAL TRIAL: NCT07356596
Title: Lower-Extremity Strength and Power in Elite Hockey Players With and Without Patellar Tendinopathy
Status: Completed | Type: Observational
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Sofia Ryman Ryman Augustsson, Associate Professor, Linnaeus University
Other Study IDs: 2025-01700-02
Record Dates: First submitted 2025-12-23; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Patellar Tendinitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unilateral PT: Ice-hockey players with unilateral patellar tendinopathy
- Bilateral PT: Ice-hockey players with bilateral patellar tendinopathy
- Control: Ice-hockey players without patellar tendinopathy

SUMMARY:
This study aims to identify differences in lower-extremity strength and power between elite ice hockey players with and without patellar tendinopathy using unilateral and bilateral comparisons. It applies a structured, cross-sectional methodology that combines clinical screening, performance testing, and ultrasound imaging to characterize patellar tendon structure and lower-limb function in elite hockey players. Players are objectively classified into healthy, unilateral, or bilateral patellar tendinopathy groups based on standardized ultrasound criteria. Strength and power outcomes are assessed under controlled conditions and normalized to body mass to allow fair between-group comparisons. Isokinetic concentric strength is evaluated during a split squat performed on a robotic resistance device, while peak power output is measured using a six-second all-out cycling test on a calibrated ergometer.

DETAILED DESCRIPTION:
This study investigates whether asymptomatic structural changes impair strength and power generation in hockey players using a between-group analysis based on patellar tendon thickness. Due to a compressed training schedule, testing occurs over consecutive days under standardized conditions. On day one, players provide informed consent and complete injury screening and anthropometric assessments. Strength and power testing is conducted on days two and three by one investigator and analyzed relative to body mass, given the association between patellar tendon thickness and BMI. On day four, a blinded investigator assesses bilateral patellar tendon thickness using ultrasound. On day five, both investigators independently analyze the images. Based on tendon thickness cutoffs, players are classified into healthy, unilateral, or bilateral tendinopathy groups, followed by between-group comparisons of strength and power outcomes.

Screening protocol: A licensed physiotherapist conducts the screening using a binary checklist (yes/no). Criteria include abnormal knee range of motion, knee pain during functional tasks, limping, positive patellar or ligament tests, joint effusion, or unilateral quadriceps atrophy (limb symmetry index <90%). Any positive finding results in immediate exclusion.

Anthropometrics: Body height and body weight are measured privately using a stadiometer and electronic scale, and body mass index is calculated.

Strength testing: Isokinetic leg strength is assessed using a split squat on a robotic resistance device at a concentric speed of 1 m/s. Players perform three maximal repetitions per leg following a standardized warm-up, and peak concentric force is recorded, with the best trial used for analysis.

Power testing: Peak power output is measured using a six-second all-out cycling test on a calibrated ergometer. After a standardized warm-up, resistance is fixed, and players sprint maximally following a countdown. Peak power output is recorded.

Ultrasound examination: Patellar tendon thickness is assessed bilaterally using ultrasound according to standardized guidelines. Players lie supine with the knee flexed ~30°, and longitudinal and transverse scans are obtained. Two independent examiners analyze images, and a tendon thickness >5 mm indicates patellar tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Elite ice-hockey player
* ≥ 18 year

Exclusion Criteria:

* injuries to lower extremity that could influence test perfomance
* deviant passive and active range of motion in the knee joint
* pain in the knee during squatting, lunging, or jumping
* limping while walking
* positive patellar The Royal London Hospital Test
* palpable or visible the knee joint effusion
* positive Lachmann, varus/valgus stress test, patellar apprehension, or Murray's/Apley's test
* hypo- or atrophic quadriceps on only one side (side difference with limb symmetry index < 90%).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty-eight male players from the Swedish Hockey League (age: 25 ± 4.6 years; body mass index: 25.5 ± 2.0) participate in this study. Based on ultrasound findings, players are classified as healthy (HG; n = 8), unilateral patellar tendinopathy (UPTG; n = 8), or bilateral patellar tendinopathy (BPTG; n = 12).
  Of 35 consenting players, only those without current or prior knee injuries affecting lower-extremity function are included. A licensed physiotherapist conducts screening, excluding five players, while two additional players are excluded due to training-related injuries.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Isokinetic leg strength | Day 2
  Isokinetic leg strength measured as the concentric peak force (Newton)
Wattbike Peak 6 test | Day 3
  A six-second "all-out" peak power test on the Wattbike measured in Watt

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT07356596/SAP_000.pdf